CLINICAL TRIAL: NCT01621685
Title: The Role of Age on the Human Cough Reflex
Brief Title: Human Safety of Capsaicin Inhalation Challenge Testing for Young and Older Men
Acronym: Capsaicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stuart M Brooks, Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IND# 69,642
Record Dates: First submitted 2010-08-05; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: COPD
Keywords: Capsaicin; Cough; Cough reflex; Inhalation agents; Inhalation challenge; TRPV1 receptor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough | interventions — Biological Products; Vaccines; Accidental Falls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spirometry, auscultation, questionnaire (Experimental): >12% fall in FEV1, wheezing on auscultation, symptom questionnaire score >4
  Interventions: Biological: biological/vaccine

INTERVENTIONS:
Biological: biological/vaccine — Inhalation studies will immediately be terminated after a significant adverse response to a particular capsaicin dose and no further testing will occur.
  Other Names: >12% fall in FEV1, wheezing on chest auscultation or >4 on Symptom Questionnaire

SUMMARY:
In 2004, the investigators initiated a human Capsaicin inhalation experiment under an Investigational New Drug (IND) protocol approved by the FDA (IND 69,642) and the subject safety procedures instituted and approved by the Institutional Review Board (IRB). As part of the study protocol, inhaled Capsaicin solutions were analyzed using high performance liquid chromatography (HPLC). The investigation employed safety procedures while conducting the human inhalation investigations. In addition, during our investigations we observed discrepancies between the predicted Capsaicin concentrations mixed by a registered pharmacist and the actual capsaicin concentrations determined by HPLC. The stability of Capsaicin solutions stored over a seven month period and refrigerated at 4degrees C and protected against ultraviolet light were examined.

DETAILED DESCRIPTION:
After a research subject's death during an inhalation study using medications/drugs not approved for this route, the FDA prohibited human use of non-approved chemicals including capsaicin administered via inhalation.

Capsaicin inhalation challenge tests (CICT) were performed on forty men of different ages utilizing pharmaceutical grade Capsaicin. Solutions were mixed by a registered pharmacist and Capsaicin doses, administered to subjects, were analyzed by high performance liquid chromatography (HPLC). Capsaicin solutions were stored in a refrigerator at 4 degrees C and shielded from ultraviolet light for 7 months. There was serial monitoring by spirometry and impulse oscillometry, electrocardiography, blood pressure, pulse and oxygen saturation measurements.

There were no adverse reactions at any dose, including the highest capsaicin concentration. Serial spirometry and impulse oscillometry, electrocardiography, blood pressure, pulse and oxygen saturation measurements did not change. The actual amount of pharmaceutical-grade capsaicin measured was 85.5% of the concentrations estimated by the registered pharmacist at time of mixing. The difference was more for the lowest 0.49 uMol dose (28.1) compared to a 2.2% lesser concentration for the 1000 uMol solution. Capsaicin concentrations fell after 3 months of storage.

Dilute capsaicin aerosol inhalation is relatively innocuous and CICT is safe. The actual amount of pharmaceutical-grade capsaicin inhaled by subjects is less than the estimate at mixing. Capsaicin loses potency after 3-months of protected storage. Inhalation studies involving non-approved drugs or chemicals/medications can be safely conducted when they follow the appropriate safety procedures such as described in this investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Men of ages 18 and 30 (Dates of birth 1973-1985) or 55-92 years old (Dates of birth 1911-1948).
2. Must not currently be a cigarette smoker. If an ex-smoker then has not smoked for at least 10 years and consumption were no more than 10 pack years.
3. Agrees to volunteers for the study and willing to sign the informed consent form.
4. There were negative/normal screening tests for the following

   1. Responses to the questionnaire deny current and prior respiratory diseases (including asthma, emphysema, chronic bronchitis, sinusitis and interstitial lung d9sase) and no current respiratory complaints (e.g., cough, wheezing, shortness of breath, allergic rhinitis, and sinusitis). Subjects must not be taking any cardiac medications or admit to a physician-diagnosed cardiac condition.
   2. "Normal" spirometry measurements with FEV1 & FVC greater than 75% predicted and FEV1/FVC more than 69%
   3. Impedance oscillometry were within normal limits
   4. "Negative" physical examination of the chest with absence of wheezing and crackles on auscultation of the chest.
   5. Exhaled nitric oxide concentration is less than 35 ppb for younger and less than 65 ppb for older groups

Exclusion Criteria:

1. men of: ages < 18, 31-54 and >92 years old;
2. current cigarette smokers or exsmokers who have smoked within the past 10 years and/or smoked more than 10 pack/years;
3. refusal to volunteer for the study and not willing to sign the informed consent form;
4. screening test not considered "normal" by physician/PI and showing one or more of the following:

   1. one or more positive response to the questionnaire(e.g., current or past respiratory diseases including asthma, emphysema, chronic bronchitis, sinusitis and interstitial lung disease; and/or; current respiratory complaints (e.g., cough, wheezing, shortness of breath, allergic rhinitis, and sinusitis) and/or; admitting to taking a cardiac medication and/or; or physician-diagnosed cardiac condition (e.g., coronary heart disease, angina, myocardial infarction, valvular heart disease, cardiomyopathy, etc.);
   2. Abnormal spirometry measurements (FEV1 &/or FVC <75% predicted and FEV1/FVC <69%);
   3. "Positive" physical examination (performed by Physician/PI) with presence of wheezing and/or crackles on auscultation of the chest;
   4. Impulse oscillometry >4 times normal limits;
   5. Exhaled nitric oxide of >35ppb for younger group and >65 ppb for older group. -

Ages: 19 Years to 92 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
>12% Fall In FEV1 | Baseline and >5 coughs 2-minutes after each inhaled capsaicin dose
  Single breaths of capsaicin were delivered in ascending order, with normal saline solution randomly interspersed to increase challenge blindness, until two (C2) and five (C5) or more coughs were reached. The different concentrations were delivered at 2 minute intervals. After each inhalation dose the following were performed: FEV1 measurement, administer of the symptom questionnaire and auscultation of the chest for wheezing.

SECONDARY OUTCOMES:
Symptom Questionnaire | Repeatedly over 1 week
  Over a 1-week period, repeated telephone calls recorded responses to 6 questions. Subjects were asked post-inhalation symptoms of: (1) heavy or difficulty in breathing; (2) phlegm production: (3) runny or irritated nose; (4) throat irritation or burning: (5) feeling of a weight or tightness of the chest; and, (6) feeling of chest burning. Any subject reporting continued symptoms of category #4 (i.e., very severe) for two or more items, compared to the baseline was asked to return for more detailed evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M. Brooks, MD, Principal Investigator — University of South Florida
Locations (1):
- College of Public Health, Tampa, Florida, United States

REFERENCES:
- [Result] Szallasi A, Blumberg P. Vanilloid (Capsaicin) Receptors and Mechanisms. Pharmacol Reviews 1999; 51:159-211 -Dicpinigaitis PV, Alva RV. Safety of capsaicin. Chest 2005; 128:196-202 -Dicpinigaitis PV. Cough reflex sensitivity in cigarette smokers. Chest 2003; 123:685-688 -Dicpinigaitis PV. Short- and long-term reproducibility of capsaicin cough challenge testing. Pulm Pharmacol Ther 2003; 16:61-65 -Broeders MEAC, Molema J, Hop WCJ, et al. Bronchial challenge, assessed with forced expiratory maneuvers and airway impedance. Respiratory Medicine 2005; 99:1046-1052 - Gordon R, Haight R, Brooks, SM.. Role of Age on Exhaled breath nitric oxide. Lung 2006 -Cortright DN, Szallas, A. Biochemical pharmacology of the vanilloid receptor TRPV1: An update. Eur. J. Biochem 1994; 271:1841-1819 -Kopec SE, DeBellis RJ, Irwin, RS. Chemical analysis of freshly prepared and stored capsaicin solutions: Implications for tussigenic challenges. Pulm Pharmacol Therapetics 2002; 15:529-534.